CLINICAL TRIAL: NCT04109391
Title: A Double-blinded Extension Study to Provide Adjuvant Treatment With Single Agent Herceptin® or TX05 and Assess Continued Safety and Immunogenicity in Subjects With HER2-positive Early Breast Cancer Following Neoadjuvant Treatment and Surgical Resection in Protocol TX05-03
Brief Title: Extension Study to Provide Adjuvant Treatment Following Neoadjuvant Treatment and Surgical Resection in Protocol TX05-03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanvex BioPharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX05-03E
Record Dates: First submitted 2019-09-20; First posted 2019-09-30 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-04

CONDITIONS: HER2-positive Breast Cancer; Early-stage Breast Cancer; Breast Cancer; Breast Neoplasms; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Test Product (TX05) (Experimental): IV trastuzumab (TX05) 8 mg/kg loading dose and then 6 mg/kg every 3 weeks for up to 13 cycles TX05 (trastuzumab): Subjects will receive up to 13 cycles of adjuvant treatment.
  These subjects received TX05 on the TX05-03 study and continued to receive TX05 in this extension study.
  Interventions: Biological: TX05 (trastuzumab)
- Reference Therapy (Herceptin) (Active Comparator): IV trastuzumab (Herceptin) TX05 8 mg/kg loading dose and then 6 mg/kg every 3 weeks for up to 13 cycles Herceptin (trastuzumab): Subjects will receive up to 13 cycles of adjuvant treatment.
  These subjects received Herceptin on the TX05-03 study and were randomized to receive Herceptin in this extension study.
  Interventions: Biological: Herceptin (trastuzumab)
- Test Product (Herceptin/TX05 Transition) (Experimental): IV trastuzumab (TX05) 8 mg/kg loading dose and then 6 mg/kg every 3 weeks for up to 13 cycles TX05 (trastuzumab): Subjects will receive up to 13 cycles of adjuvant treatment.
  These subjects received Herceptin on the TX05-03 study and were randomized to receive TX05 in this extension study.
  Interventions: Biological: TX05 (trastuzumab)

INTERVENTIONS:
Biological: TX05 (trastuzumab) — Subjects will receive up to 13 cycles of adjuvant treatment.
  Arms: Test Product (Herceptin/TX05 Transition); Test Product (TX05)
Biological: Herceptin (trastuzumab) — Subjects will receive up to 13 cycles of adjuvant treatment.
  Arms: Reference Therapy (Herceptin)

SUMMARY:
This is an extension study to provide adjuvant treatment with single agent Herceptin or TX05 and assess continued safety and immunogenicity in subjects with HER2-positive early breast cancer following neoadjuvant treatment and surgical resection in Protocol TX05-03.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Females ≥ 18 years of age.
* Completed neoadjuvant treatment (regardless of treatment arm) in the TX05/ Herceptin neoadjuvant study and the investigator believes the subject requires continued access to single agent trastuzumab in order to continue deriving clinical benefit.
* Successfully undergone surgical resection of their primary tumor with no evidence of residual disease (as determined by local assessment) and no other adjuvant therapy, other than trastuzumab, is planned. However, subjects will be allowed to receive hormonal therapy if they have hormone receptor positive tumors. Subjects will also be allowed to receive adjuvant radiation therapy, if required by their treating physician.
* Able to comply with the study protocol.
* Female subjects of childbearing potential must have a negative serum pregnancy test within 14 days of first administration of study drug and agree to use effective contraception (hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide) throughout the study period and for 7 months after last administration of study drug.

Exclusion Criteria:

* Breast cancer metastases or residual disease post operatively (as determined by local assessment).
* History or presence of a medical condition or disease that in the investigator's opinion would place the subject at an unacceptable risk for study participation.
* Lactating or pregnant female.
* Women of childbearing potential who do not consent to use highly effective methods of birth control (e.g. true abstinence [periodic abstinence {e.g. calendar ovulation, symptothermal, post-ovulation methods} and withdrawal are not acceptable methods of contraception], sterilization, or other non-hormonal forms of contraception) during treatment and for at least 7 months after the last administration of study drug. Subjects must agree to not breast-feed while receiving study drug.
* Any condition that in the opinion of the Investigator represents an obstacle for study conduct and/or represents a potential unacceptable risk for subjects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Mills, PhD, Study Director — Tanvex BioPharma USA, Inc.
Locations (86):
- Belarus (6):
  - Tanvex Investigational Site 1006E, Grodno
  - Tanvex Investigational Site 1003E, Homyel
  - Tanvex Investigational Site 1008E, Lesnoy
  - Tanvex Investigational Site 1002E, Minsk
  - Tanvex Investigational Site 1005E, Mogilev
  - Tanvex Investigational Site 1001E, Vitebsk
- Chile (2):
  - Tanvex Investigational Site 4001E, Temuco
  - Tanvex Investigational Site 4002E, Viña del Mar
- Georgia (6):
  - Tanvex Investigational Site 5006E, Batumi
  - Tanvex Investigational Site 5002E, Batumi
  - Tanvex Investigational Site 5001E, Tbilisi
  - Tanvex Investigational Site 5005E, Tbilisi
  - Tanvex Investigational Site 5010E, Tbilisi
  - Tanvex Investigational Site 5008E, Tbilisi
- Tanvex Investigational Site 6003E, Budapest, Hungary
- India (10):
  - Tanvex Investigational Site 7031E, Nashik, Maharashtra
  - Tanvex Investigational Site 7033E, Ahmedabad
  - Tanvex Investigational Site 7019E, Bangalore
  - Tanvex Investigational Site 7022E, Belagavi
  - Tanvex Investigational Site 7045E, Hyderabad
  - Tanvex Investigational Site 7036E, Hyderabad
  - Tanvex Investigational Site 7006E, Kolkata
  - Tanvex Investigational Site 7001E, Nashik
  - Tanvex Investigational Site 7015E, Pune
  - Tanvex Investigational Site 7017E, Vijayawada
- Mexico (5):
  - Tanvex Investigational Site 2109E, Aguascalientes
  - Tanvex Investigational Site 2103E, Monterrey
  - Tanvex Investigational Site 2106E, Oaxaca City
  - Tanvex Investigational Site 2110E, Tequisquiapan
  - Tanvex Investigational Site 2108E, Zapopan
- Peru (9):
  - Tanvex Investigational Site 1101E, Arequipa
  - Tanvex Investigational Site 1107E, Arequipa
  - Tanvex Investigational Site 1104E, Chiclayo
  - Tanvex Investigational Site 1105E, Lima
  - Tanvex Investigational Site 1112E, Lima Cercado
  - Tanvex Investigational Site 1108E, San Borja
  - Tanvex Investigational Site 1102E, San Isidro
  - Tanvex Investigational Site 1109E, Surquillo
  - Tanvex Investigational Site 1103E, Trujillo
- Philippines (6):
  - Tanvex Investigational Site 1211E, Cebu City
  - Tanvex Investigational Site 1212E, Davao City
  - Tanvex Investigational Site 1214E, Makati City
  - Tanvex Investigational Site 1209E, Quezon City
  - Tanvex Investigational Site 1213E, Quezon City
  - Tanvex Invesitgational Site 1210E, Santo Tomas
- Russia (24):
  - Tanvex Investigational Site 1513E, Sochi, Krasnodarskiy Kray
  - Tanvex Investigational Site 1535E, Arkhangelsk
  - Tanvex Investigational Site 1531E, Belgorod
  - Tanvex Investigational Site 1502E, Kaluga
  - Tanvex Investigational Site 1505E, Kislino
  - Tanvex Investigational Site 1529E, Krasnodar
  - Tanvex Investigational Site 1512E, Krasnoyarsk
  - Tanvex Investigational Site 1530E, Moscow
  - Tanvex Investigational Site 1507E, Moscow
  - Tanvex Investigational Site 1511E, Novosibirsk
  - Tanvex Investigational Site 1503E, Omsk
  - Tanvex Investigational Site 1509E, Omsk
  - Tanvex Investigational Site 1537E, Orenburg
  - Tanvex Investigational Site 1526E, Pesochnyy
  - Tanvex Investigational Site 1510E, Pushkin
  - Tanvex Investigational Site 1521E, Rostov-on-Don
  - Tanvex Investigational Site 1516E, Saint Petersburg
  - Tanvex Investigational Site 1523E, Saint Petersburg
  - Tanvex Investigational Site 1524E, Saint Petersburg
  - Tanvex Investigational Site 1525E, Saint Petersburg
  - Tanvex Investigational Site 1506E, Saint Petersburg
  - Tanvex Investigational Site 1501E, Saint Petersburg
  - Tanvex Investigational Site 1508E, Saransk
  - Tanvex Investigational Site 1534E, Yaroslavl
- Ukraine (17):
  - Tanvex Investigational Site 1820E, Antonivka
  - Tanvex Investigational Site 1803E, Chernihiv
  - Tanvex Investigational Site 1808E, Chernihiv
  - Tanvex Investigational Site 1821E, Chernivtsi
  - Tanvex Investigational Site 1824E, Dnipro
  - Tanvex Investigational Site 1811E, Kiev
  - Tanvex Investigational Site 1802E, Kiev
  - Tanvex Investigational Site 1819E, Kropyvnytskyi
  - Tanvex Investigational Site 1814E, Kropyvnytskyi
  - Tanvex Investigational Site 1804E, Kryvyi Rih
  - Tanvex Investigational Site 1815E, Kyiv
  - Tanvex Investigational Site 1809E, Kyiv
  - Tanvex Investigational Site 1810E, Odesa
  - Tanvex Investigational Site 1806E, Sumy
  - Tanvex Investigational Site 1822E, Ternopil
  - Tanvex Investigational Site 1818E, Vinnytsia
  - Tanvex Investigational Site 1813E, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product (TX05 Only): IV trastuzumab (TX05) 8 mg/kg loading dose and then 6 mg/kg every 3 weeks for up to 13 cycles
  TX05 (trastuzumab): Subjects will receive up to 13 cycles of adjuvant treatment.
  These subjects received TX05 on the TX05-03 study and continued to receive TX05 in this extension study.
- Reference Therapy (Herceptin Only): IV trastuzumab (Herceptin) TX05 8 mg/kg loading dose and then 6 mg/kg every 3 weeks for up to 13 cycles
  Herceptin (trastuzumab): Subjects will receive up to 13 cycles of adjuvant treatment.
  These subjects received Herceptin on the TX05-03 study and continued to receive Herceptin in this extension study.
Period: Overall Study
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition)
Started | 175 | 82 | 81
Completed | 165 | 77 | 77
Not Completed | 10 | 5 | 4
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Subject refused to continue, AE and 2 patients only received 10 of 13 cycles | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition) | Total
Number analyzed (Participants) | 175 | 82 | 81 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.43) | 53.7 (10.12) | 54.0 (10.71) | 54.6 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 82 | 81 | 338
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 12 | 10 | 51
  Not Hispanic or Latino | 146 | 70 | 71 | 287
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 2 | 8
  Asian | 23 | 13 | 17 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 136 | 64 | 57 | 257
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 4 | 5 | 20
Hormone Receptor Status [Count of Participants; unit: Participants]
  Positive | 100 | 50 | 48 | 198
  Negative | 75 | 32 | 33 | 140
Tumor Stage [Count of Participants; unit: Participants] — Enrolled subjects should have Stage II/IIIabreast cancer.
  Stage will be determined by the American Joint Committee onCancer (AJCC) TNM (tumor size, lymph node involvement,metastasis to distant sites) staging system.
  A low grade number (grade 1) usually means the cancer isslower-growing and less likely to spread. A high grade number(grade 3) means a faster-growing cancer that's more likely tospread. An intermediate grade number (grade 2) means thecancer is growing faster than a grade 1 cancer but slower than agrade 3 cancer.
  Participants
    Stage IIa | 65 | 28 | 32 | 125
    Stage IIb | 78 | 41 | 35 | 154
    Stage IIIa | 32 | 13 | 14 | 59
ECOG [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease activities without restriction
  Grade 1: Restricted in physically strenuous activity but ambulatory andable to carry out work of a light or sedentary nature.
  Grade 2: Ambulatory and capable of all self-care but unable to carryout any work activities. Up and about more than 50% of waking hours.
  Grade 3: Capable of only limited self-care, confined to bed or chairmore than 50% of waking hours.
  Grade 4: Completely disabled. Cannot carry on any self-care. Totallyconfined to bed or chair.
  Grade 5: Dead
  Participants
    Grade 0 | 142 | 56 | 64 | 262
    Grade 1 | 29 | 24 | 16 | 69
    Grade 2 | 0 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0 | 0
    Missing | 4 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Assessments (ADA and Nab)
Description: Samples for the evaluation of anti-drug antibodies (ADA), including neutralizing antibodies (Nab) were obtained before the administration of Cycle 1 (Week 0), Cycle 6 (Week 15), and the EOT/ET Visit. Only subjects with a positive ADA result were further tested for ADA cross-reactivity and Nab. Only subjects with a positive Nab result were further tested for Nab cross-reactivity.
Time Frame: Assessed from first infusion through end of treatment (Week 45) or Early Termination visit. Each cycle is 3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition)
Number analyzed (Participants) | 175 | 82 | 81
Participants
  Baseline: ADA Positive | 3 | 2 | 3
  Baseline: Nab Positive | 0 | 0 | 0
  Baseline: ADA Negative | 159 | 77 | 74
  Baseline: Not evaluated | 13 | 3 | 4
  Cycle 6 Week 15: ADA Positive | 1 | 1 | 4
  Cycle 6 Week 15: Nab Positive | 0 | 0 | 0
  Cycle 6 Week 15: ADA Negative | 164 | 74 | 74
  Cycle 6 Week 15: Not evaluated | 10 | 7 | 3
  End of Study/Early Terminiation: ADA Positive | 4 | 1 | 2
  End of Study/Early Terminiation: Nab Positive | 0 | 0 | 0
  End of Study/Early Terminiation: ADA Negative | 146 | 75 | 71
  End of Study/Early Terminiation: Not evaluated | 25 | 6 | 8

2. Primary Outcome: Disease-Free Survival
Description: DFS, defined as the time from randomization in the neoadjuvant study (Protocol TX05-03) to the documentation of a first failure, where a failure was the recurrence of breast cancer or a diagnosis of a second primary cancer.
Time Frame: Through study completion/end of treatment (Week 45).
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition)
Number analyzed (Participants) | 175 | 82 | 81
Participants
  Recurrence of Breast Cancer or a Diagnosis of a Second Primary Cancer | 6 | 5 | 3
  No recurrence of Breast Cancer and No Diagnosis of a Second Primary Cancer | 160 | 73 | 76
  Discontinued form Study | 8 | 4 | 2
  No Post Baseline or No Evaluable Post Baseline | 1 | 0 | 0
  No Baseline or No Evaluable Baseline Assessment | 0 | 0 | 0
  Death | 0 | 0 | 0

3. Primary Outcome: Overall Survival
Description: OS, defined as the time from randomization in the neoadjuvant study (Protocol TX05-03) until death from any cause.
Time Frame: Through study completion/end of treatment (Week 45).
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition)
Number analyzed (Participants) | 175 | 82 | 81
Participants
  Last known alive | 175 | 82 | 80
  Lost to Follow-Up | 0 | 0 | 0
  Death | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from Day 1 (Week 0) of Cycle 1 of study treatment through End of Treatment (Week 45), with the exception of any ongoing study drug-related AEs, which were to be followed until the event was resolved, considered stable, or the investigator determined the AE was no longer clinically significant.
Description: Ongoing drug-related AEs and SAEs from the neoadjuvant study (Protocol TX05-03) and any SAEs that occurred after completion of the neoadjuvant study were recorded at Screening in the subject's medical history, while AEs occurring in this extension study were recorded from Day 1 (Week 0) of Cycle 1 of study treatment.
Arm/Group | Test Product (TX05 Only) | Reference Therapy (Herceptin Only) | Test Product (Herceptin/TX05 Transition)
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/82 | 1/81
Serious Adverse Events (participants affected / at risk) | 4/175 | 3/82 | 2/81
Other Adverse Events (participants affected / at risk) | 49/175 | 15/82 | 15/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (TX05 Only) (N=175) | Reference Therapy (Herceptin Only) (N=82) | Test Product (Herceptin/TX05 Transition) (N=81)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection/ (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture/ (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (TX05 Only) (N=175) | Reference Therapy (Herceptin Only) (N=82) | Test Product (Herceptin/TX05 Transition) (N=81)
Respiratory Tract Infection (Infections and infestations) | 6 (6) | 2 (2) | 5 (5)
Alanine Aminotransferase Increased (Investigations) | 10 (11) | 2 (6) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 9 (10) | 1 (3) | 3 (3)
Headache (Nervous system disorders) | 9 (13) | 5 (8) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 2 (2)
Asthenia (General disorders) | 10 (12) | 4 (4) | 3 (4)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 13 (13) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04109391/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04109391/SAP_001.pdf